CLINICAL TRIAL: NCT05135403
Title: ASSURE WCD Clinical Evaluation - Post Approval Study (ACE-PAS)
Acronym: ACE-PAS
Status: Recruiting | Type: Observational
Sponsor: Kestra Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-00187-01
Record Dates: First submitted 2021-08-30; First posted 2021-11-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ASSURE Registry Patients: Patient prescribed the ASSURE WCD who have also consented to participate in the ASSURE Patient Registry. Patients include those with reduced left ventricular ejection fraction (LVEF) and recent myocardial infarction, recent coronary revascularization, or new onset heart failure (HF) to allow for optimization of medical therapy and re-evaluation of cardiac function. Additional indications include ICD explant due to infection, postponed ICD implant, and pending heart transplant.
  Interventions: Device: Defibrillation

INTERVENTIONS:
Device: Defibrillation — External defibrillation from a wearable cardioverter defibrillator

SUMMARY:
Active surveillance study using real-world data collected in the ASSURE Patient Registry. Outcome measures are based on analysis of ASSURE Registry data including data recorded by the WCD then annotated by clinical experts in electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient prescribed the ASSURE wearable cardioverter defibrillator
* Provided written informed consent to participate in the ASSURE Patient Registry

Exclusion Criteria:

* Patients who do not meet the Inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The ASSURE Wearable Cardioverter Defibrillator (WCD) system is indicated for adult patients who are at risk or at perceived risk of sudden cardiac arrest (SCA) and are not immediate candidates for, or refuse, an implantable defibrillator.
Sampling Method: Probability Sample
Enrollment: 5179 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall shock conversion rate | Up to 3 years
  Percent of spontaneous episodes of ventricular tachycardia/ventricular fibrillation (VT/VF) successfully converted with one or more shocks ≥ 89.0%
Inappropriate shocks per patient month | Up to 3 years
  Total inappropriate shocks/cumulative months of WCD use for all patients ≤ 0.0075

SECONDARY OUTCOMES:
First shock conversion rate | Up to 3 years
  Percent of spontaneous episodes of ventricular tachycardia/ventricular fibrillation (VT/VF) converted with a single shock. (report only)
Inappropriate shock rate | Up to 3 years
  Percent of patients who experience at least one inappropriate shock (report only)

OTHER OUTCOMES:
Appropriate shock rate per month | Up to 3 years
  Number of appropriate shocks/cumulative months of WCD use
Appropriate shock rate | Up to 3 years
  Percent of patients who experience at least one appropriate shock
Total Shocks delivered | Up to 3 years
  Number of shocks delivered
Shocks diverted | Up to 3 years
  Number of shocks diverted by patients
False positive shock alarm rate | Up to 3 years
  Number of false positive shock alarms/cumulative WCD use
True positive shock alarm rate | Up to 3 years
  Number of true positive shock alarms/cumulative WCD use
Adverse events | Up to 3 years
  Adverse events related to use of the WCD
Average daily device use | Up to 3 years
  Average daily use of the WCD in hours per day
Cumulative device use | Up to 3 years
  Cumulative device use in days

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Poole, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No